CLINICAL TRIAL: NCT04275089
Title: Early Feasibility Prospective Open-Label Study to Assess the Function of a Novel Pessary for the Non-Surgical Management of Pelvic Organ Prolapse
Brief Title: Early Feasibility Study of the Reia Vaginal Pessary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-001
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: Pelvic Organ Prolapse; Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Reia Vaginal Pessary (Experimental)
  Interventions: Device: Reia Vaginal Pessary

INTERVENTIONS:
Device: Reia Vaginal Pessary — Reia Vaginal Pessary

SUMMARY:
This is an early feasibility open-label non-randomized trial to obtain preliminary information about the function and effectiveness of a novel vaginal pessary for the use in women who suffer from symptoms of pelvic organ prolapse (POP). Recruited patients will have Stage II POP or greater and will be current users of a legally marketed vaginal pessary. In a single visit, data will be collected on the performance and comfort of the subject's current pessary. After placement of a study pessary, comparative data will be collected between subject's current pessary and the study pessary on ability to support prolapse. The study pessary's function will be assessed under controlled circumstances. The patient will have her current pessary replaced at the conclusion of the visit. Results will be used to inform future design modifications of the study pessary.

ELIGIBILITY:
Inclusion Criteria:

* Women with Stage II pelvic organ prolapse or greater
* Current ring style or Gellhorn pessary users inclusive of sizes 1.5"-3.5"
* Capable of giving informed consent

Exclusion Criteria:

* Pregnancy
* Deep vaginal erosion noted with removal of current pessary
* Presence of vesicovaginal fistula
* Presence of rectovaginal fistula
* Vaginal, rectal, or bladder tumor
* Inflammatory Bowel Disease
* Presence of open wound or tear near vagina or anus by exam prior to removal of current pessary
* Current vaginal or urinary infection requiring treatment
* Previous pelvic floor surgery in last 12 months
* Congenital malformation of bladder, rectum, or vagina
* Significant medical condition interfering with study participation (psychologic, neurologic, active drug/alcohol abuse, etc.)
* Planning pregnancy in next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Strohbehn, MD, Principal Investigator — Dartmouth-Hitchcock Clinic
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reia Vaginal Pessary
Started | 15
Completed | 14
Not Completed | 1
Not completed — Unable to be fit with Reia pessary | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 78 [63 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Pessary type [Count of Participants; unit: Participants]
  Gellhorn | 8
  Ring | 7
BMI [Count of Participants; unit: Participants]
  <20 | 1
  20-30 | 9
  >30 | 5
Menopause status [Count of Participants; unit: Participants]
  Post menopause | 15
  Pre menopause | 0
Prolapse severity [Count of Participants; unit: Participants] — POP-Q Stage - higher is worse. Prolapse stage recorded from chart abstraction from most recent clinical evaluation of prolapse stage.
  Participants
    Stage II | 8
    Stage III | 5
    Stage IV | 2

OUTCOME MEASURES:

1. Primary Outcome: The Ability of the Study Device to be Retained During Valsalva Compared to the Ability of the Subject's Current Pessary to be Retained During Valsalva (Change in Distance Between Current Pessary and Study Pessary to Leading Edge to the Hymen)
Description: The subject will be asked to Valsalva with their current pessary in place, and the distance from the leading edge of the current pessary to the hymen will be measured in centimeters. After the current pessary is removed and with the study pessary in place, the subject will be asked to Valsalva again. The distance from the leading edge of the study pessary to the hymen will be measured in centimeters. In order to assess the ability of the study pessary to function and be retained, the measurements will be compared.
Time Frame: During treatment - within 1 hour
Measure: Median (Standard Deviation); unit: cm
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 14
cm | 0 (1.7)

2. Primary Outcome: The Ability of the Study Device to be Retained Throughout Regular Activity (by Vaginal Examination)
Description: With the study pessary in place, the subject will be asked to ambulate for 10 minutes and attempt to void. Following these activities, whether the pessary was retained or expelled will be recorded.
Time Frame: During treatment - within 1 hour
Measure: Number; unit: participants
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 14
participants
  pessary retained | 14
  pessary expelled | 0

3. Secondary Outcome: Shape of the Study Pessary During Expulsion if it is Not Able to be Retained (by Vaginal Examination)
Description: The subject will be asked to Valsalva. If the study device is expelled during Valsalva, whether the study device was expelled fully deployed or whether it prematurely folded to its collapsed state will be recorded.
Time Frame: During treatment - within 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 14
Participants
  Not expelled | 14
  Expelled in collapsed state | 0
  Expelled in deployed state | 0

4. Secondary Outcome: Orientation of the Study Pessary Stem Following Regular Activity (by Vaginal Examination)
Description: Following ambulation and attempting to void and prior to removing the study pessary, it will be recorded if the study device's stem rotated out of its original inserted position.
Time Frame: During treatment - within 1 hour
Measure: Number; unit: participants
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 14
participants
  Rotated | 1
  Not rotated | 13

5. Secondary Outcome: Discomfort Experienced With Removal of the Study Pessary Subtracted From the Discomfort Experienced With Removal of the Subject's Current Pessary (Change in VAS) [Positive Score Indicates Lower Discomfort With Study Pessary]
Description: To indicate discomfort, the subject will be shown and asked to mark a visual analogue scale (VAS) after removal of her current pessary and before using the study pessary. The VAS will be a 10 centimeter linear continuum in which 0 represents no pain and 10 represents worst pain. After use of the study pessary and upon removal of the study pessary, the subject will be shown and asked to mark another VAS. In order to assess the discomfort experienced during removal of the study pessary, the distance from 0 to the subject's mark will be measured and compared between the two scales. The outcome measure is [VAS after removal of current pessary] - [VAS after removal of study pessary].
Time Frame: During treatment - within 1 hour
Population: 1 subject arrived without current pessary in place, so no current pessary VAS removal score was recorded.
Measure: Mean (Inter-Quartile Range); unit: cm
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 13
cm | 1.4 [-1.3 to 4.3]

6. Secondary Outcome: Discomfort Experienced With Insertion of the Study Pessary Subtracted From the Discomfort Experienced With Insertion of the Subject's Current Pessary (Change in VAS) [Positive Score Indicates Lower Discomfort With Study Pessary]
Description: To indicate discomfort, the subject will be shown and asked to mark a VAS after insertion of the study pessary. The VAS will be a 10 centimeter linear continuum in which 0 represents no pain and 10 represents worst pain. After use of the study pessary and upon insertion of the subject's current pessary, the subject will also be shown and asked to mark another VAS. In order to assess the discomfort experienced during insertion of the study pessary, the distance from 0 to the subject's mark will be measured and compared between the two scales. The outcome measure is [VAS after insertion of current pessary] - [VAS after insertion of study pessary].
Time Frame: During treatment - within 1 hour
Population: 1 subject did not have current pessary reinserted due to discomfort with insertion of the current pessary.
Measure: Mean (Inter-Quartile Range); unit: cm
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 13
cm | 1.3 [-1.2 to 5.7]

7. Secondary Outcome: Global Comfort Associated With Use of the Study Pessary (by Verbal Description)
Description: Following insertion of the subject's current pessary, and after the subject is dressed, she will be asked whether the study pessary was more, less, or as comfortable as her current pessary when it was in situ. If she responds it was more or less comfortable, she will be asked to describe why.
Time Frame: Post treatment - within or at 1 hour
Population: Data was not collected by the study team for 1 subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Reia Vaginal Pessary
Number analyzed (Participants) | 13
Participants
  Study pessary more comfortable | 2
  Equal comfort | 6
  Current pessary more comfortable | 5

ADVERSE EVENTS:
Time Frame: Duration of subject's sole study visit - within one hour
Arm/Group | Reia Vaginal Pessary
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT04275089/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04275089/SAP_001.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04275089/ICF_002.pdf